CLINICAL TRIAL: NCT05856851
Title: Intra-arterial Alteplase for Acute Ischemic Stroke After Mechanical Thrombectomy (PEARL): A Multicenter, Prospective, Open-label, Blinded Endpoint, Randomized Controlled Trial
Brief Title: Intra-arterial Alteplase for Acute Ischemic Stroke After Mechanical Thrombectomy
Acronym: PEARL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2023-390-02
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-arterial alteplase (Experimental): Participants in the experimental group will receive a 15-minute continuous infusion of intra-arterial alteplase at a drug concentration of 1.0 mg/ml. 15 minutes after the start of intra-arterial thrombolysis, the infusion will be stopped and an angiogram will be performed to assess the eTICI score. If the angiographic eTICI score improves from the baseline score, the procedure will be terminated, otherwise, a new angiogram will be repeated 5-10 minutes after the end of drug administration.
  Interventions: Drug: Alteplase
- Standard medical treatment (No Intervention): Participants allocated to the control group will receive standard medical treatment without intra-arterial alteplase after mechanical thrombectomy.

INTERVENTIONS:
Drug: Alteplase — See arm/group descriptions.
  Other Names: Intra-arterial alteplase after mechanical thrombectomy
  Arms: Intra-arterial alteplase

SUMMARY:
A multicenter, prospective, open-label, blinded endpoint, randomized controlled trial aiming at evaluating the efficacy and safety of intra-arterial recombinant human tissue plasminogen activator (rt-PA) after successful recanalization of acute large vessel occlusion in the anterior circulation by mechanical thrombectomy in improving the 90-day functional outcome.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, open-label, blinded endpoint, randomized controlled trial designed to evaluate the efficacy and safety of intra-arterial recombinant human tissue plasminogen activator (rt-PA) after successful recanalization of acute large vessel occlusion in the anterior circulation by mechanical thrombectomy (eTICI 2b50/3). The primary outcome is the proportion of patients with a 90-day modified Rankin scale (mRS) of 0-1.

Study intervention: (1) Participants in the experimental group will receive intra-arterial alteplase (a dose of 0.225 mg/kg and a maximum dose of 20 mg) after the mechanical thrombectomy, and will receive standard medical treatment after the procedure. (2) Participants in the control group will receive standard medical treatment without intra-arterial alteplase.

A total of 324 participants are anticipated to be recruited for this study, with 162 participants in each group (1:1 ratio).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Clinical diagnosis of acute ischemic stroke.
3. Time from symptom onset to randomization within 24 hours, including wake-up stroke or no-witness stroke; the onset time refers to "Last Known Well" (LKW).
4. CTA or MRA confirmed occlusion of the intracranial segment of the internal carotid artery, or M1 or M2 segment of the middle cerebral artery; stable eTICI score of 2b50-3 after mechanical thrombectomy, with or without intravenous thrombolysis. Patients with an eTICI score of 2b50-3 on the diagnostic cerebral angiography before mechanical thrombectomy are also eligible for the study.
5. Baseline NIHSS of 6-25.
6. NCCT/DWI-MRI ASPECTS ≥ 6;
7. Pre-stroke mRS score ≤ 1, or mRS >1 but not related to neurological disease (e.g., amputation, blindness).
8. Signed informed consent.

Exclusion Criteria:

1. Contraindication to rt-PA (except time to therapy).
2. Planned use of dual antiplatelet therapy within the first 24 hours after mechanical thrombectomy.
3. Angiographic evaluation showing dissection, severe stenosis, or complete occlusion of the carotid artery, which requires the use of carotid artery stents during the endovascular procedure.
4. Suspected cerebral vasculitis based on medical history and/or angiographic evaluation.
5. Women who are pregnant or breastfeeding.
6. Participation in other clinical trials.
7. Preoperative intracranial hemorrhage confirmed by cranial CT or MRI.
8. Known genetic or acquired bleeding disposition with anticoagulation factor deficiency.
9. Coagulation disorder with INR > 1.7 or use of new oral anticoagulants (within 48 hours of symptom onset).
10. Platelet count <50X10^9/L.
11. Suspected vascular occlusion as a result of infective endocarditis.
12. Known severe renal insufficiency with glomerular filtration rate <30 ml/min or blood creatinine >220 μmol/L (2.5 mg/dl).
13. Severe allergy to contrast (non-mild rash allergy) or absolute contraindication to iodine contrast.
14. Suspected aortic dissection.
15. Previous parenchymal organ surgery or biopsy in the last 1 month;
16. Any active bleeding or recent bleeding (gastrointestinal, urinary tract bleeding, etc.) in the last 1 month;
17. SBP > 185 mmHg or DBP > 110 mmHg refractory to treatment.
18. Anticipated life expectancy < 6 months (e.g., malignancy, severe cardiopulmonary disease, etc.).
19. Any condition that, in the judgment of the investigator, makes the patient unsuitable for this study or where this study may impose a significant risk to the patient (e.g., inability to understand and/or comply with study procedures and/or follow-up due to psychiatric disorders, cognitive or emotional impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale score (mRS) 0-1 | 90(±7) days
  The proportion of the modified Rankin Scale score (mRS) 0-1 at 90 days.

SECONDARY OUTCOMES:
Change of infarct volume from baseline | 7(±1) days
  The change of infarct volume at 7(±1) days or discharge (whichever occurred first) on non-contrast CT, or at 48(±12) hours on MRI
The volume of Tmax>6s on CTP | 24(±12) hours
  The volume of Tmax>6s on CTP at 24(±12) hours
The shift analysis of the modified Rankin Scale (mRS) | 90(±7) days
  The shift analysis of the modified Rankin Scale (mRS) at 90 days
The modified Rankin Scale score (mRS) 0-2 | 90(±7) days
  The proportion of the modified Rankin Scale score (mRS) 0-2 at 90 days.
The modified Rankin Scale score (mRS) 0-3 | 90(±7) days
  The proportion of the modified Rankin Scale score (mRS) 0-3 at 90 days.
The proportion of NIHSS 0-1 or ≥10 points reduction | 48 (±12) hours
  The proportion of NIHSS 0-1 or ≥10 points reduction at 48 (±12) hours
Quality of Life (EQ-5D-5L) | 90(±7) days
  The value of Quality of Life (EQ-5D-5L) at 90 days

OTHER OUTCOMES:
SAFETY OUTCOME: Symptomatic intracranial hemorrhage | 24 (±12) hours
  Symptomatic intracranial hemorrhage within 36 hours (according to Heidelberg criteria)
SAFETY OUTCOME: Mortality | 90(±7) days
  Mortality at 90 days
SAFETY OUTCOME: Any intracranial hemorrhage | 24 (±12) hours
  Any intracranial hemorrhage within 36 hours (according to Heidelberg criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Yajie Liu, Principal Investigator — Shenzhen Hospital of Southern Medical University
Locations (2):
- China (2):
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available from Principal Investigators (Prof. Yamei Tang and Prof. Yajie Liu) upon reasonable request 6 months after the trial completion.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the trial completion.
Access Criteria: The IPD will be available from Principal Investigators (Prof. Yamei Tang and Prof. Yajie Liu) upon reasonable request.

REFERENCES:
- [Derived] Yang X, He X, Pan D, Xu Y, Peng H, Li K, Zhang M, Zhu Y, Chen Y, He B, Zhou H, Li J, Hou H, Sun H, Liu Y, Tang Y. Intra-arterial alteplase for acute ischaemic stroke after mechanical thrombectomy (PEARL): rationale and design of a multicentre, prospective, open-label, blinded-endpoint, randomised controlled trial. BMJ Open. 2024 Nov 5;14(11):e091059. doi: 10.1136/bmjopen-2024-091059. PMID 39500603